CLINICAL TRIAL: NCT03657160
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Vedolizumab in the Prophylaxis of Intestinal Acute Graft Versus-Host Disease in Subjects Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Vedolizumab in the Prophylaxis of Intestinal Acute Graft Versus Host Disease (aGVHD) in Participants Undergoing Allogeneic Hematopoietic Stem Cell (Allo-HSCT) Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Vedolizumab-3035; 2018-002141-11 (EudraCT Number); JapicCTI-184221 (Registry Identifier: JapicCTI); U1111-1216-2319 (Registry Identifier: WHO)
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Hematopoietic Stem Cells
Keywords: Drug Therapy
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Vedolizumab placebo-matching, intravenous (IV) infusion, once on Day -1 along with background graft-versus-host disease (GvHD) prophylaxis regimen prior to Allo-HSCT and once on Days +13, +41, +69, +97, +125, and +153 post Allo-HSCT up to the end of study treatment (up to 182 days).
  Interventions: Drug: Vedolizumab Placebo
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once on Day -1 along with background GvHD prophylaxis regimen prior to Allo-HSCT and once on Days +13, +41, +69, +97, +125, and +153 post Allo-HSCT up to the end of study treatment (up to 182 days).
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab Placebo — Vedolizumab placebo-matching IV infusion.
  Arms: Placebo
Drug: Vedolizumab — Vedolizumab IV infusion.
  Other Names: MLN0002
  Arms: Vedolizumab 300 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of vedolizumab when added to background aGvHD prophylaxis regimen compared to placebo and background aGvHD prophylaxis regimen on intestinal aGvHD-free survival by Day +180 in participants who receive allo-HSCT as treatment for a hematologic malignancy or myeloproliferative disorder.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who are undergoing allo-HSCT transplantation. This study will look at the efficacy and safety of vedolizumab in the prophylaxis of intestinal aGvHD in participants undergoing allo-HSCT transplantation.

The study will enroll approximately 558 participants. Participants will be randomly assigned (by chance, like flipping a coin) in 1:1 ratio to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need) along with background GvHD prophylaxis regimen:

* Vedolizumab 300 mg
* Placebo (dummy inactive intravenous infusion)

This multi-center trial will be conducted Worldwide. The overall time to participate in this study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Must be >= 18 years of age and, in selected countries, adolescents aged 12 years and greater and weighing >=30 kilogram (kg) at time of randomization.
2. Must undergo deoxyribose nucleic acid (DNA)-based human leukocyte antigen (HLA) matching and be 8 of 8 or 7 of 8 HLA-matched (singe allele or antigen mismatch at HLA-A, -B, and -C, and HLA-DRB1 is allowable) unrelated hematopoietic stem cell transplantation (HSCT) from either peripheral blood or bone marrow stem cells for a hematologic malignancy or myeloproliferative disorder.
3. For whom a myeloablative conditioning or reduced intensity conditioning (RIC) is planned.
4. Allo-HSCT eligible (meeting institutional criteria)-participants planned medical care should include aGvHD prophylaxis with a combination of calcineurin inhibitor (CNI) (cyclosporine [CYS] or tacrolimus [TAC]) and methotrexate (MTX) or CNI and mycophenolate mofetil (MMF). With the exception of antithymocyte globulin (ATG) (antithymocyte globulin-Fresenius [ATG-F] or thymoglobulin), all other therapies, approved or investigational, for GvHD prophylaxis are excluded.
5. Eastern Cooperative Oncology Group (ECOG) performance status of <= 2 for participants aged >=18 years at randomization or >=60 % using the Karnofsky performance status for adolescent participants aged >=16 years at randomization or the Lansky performance status for adolescent participants aged 12 to < 16 years at randomization.

Exclusion Criteria:

1. Had prior allo- HSCT.
2. Planned umbilical cord blood transplant or planned to receive posttransplant cyclophosphamide, in vivo or ex vivo T cell-depleted hematopoietic stem cells (HSCs) with the exception of ATG (ATG-F or thymoglobulin).
3. Planned allo-HSCT for nonmalignant hematological disorders (example, aplastic anemia, sickle cell anemia, thalassemias, Fanconi anemia or immunodeficiency).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (139):
- United States (27):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - David Geffen School of Medicine at University of California Los Angeles, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center - The Columbia Center for Translational Immunology, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Massey Cancer Center, Richmond, Virginia
- Argentina (3):
  - Fundacion Favaloro Hospital Universitario, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- Australia (5):
  - Saint Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Austin Health, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Ordensklinikum Linz Elisabethinen, Linz, Upper Austria, Austria
- Belgium (2):
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Ziekenhuisnetwerk Stuivenberg, Antwerp
- Brazil (7):
  - Hospital Universitario Walter Cantidio - Universidade Federal do Ceara, Fortaleza, Ceará
  - Instituto do Cancer e Transplante de Curitiba, Curitiba, Paraná
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente - A.C.Camargo Cancer Center, São Paulo
  - Instituto Brasileiro de Controle do Cancer - Sao Camilo Oncolgia, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saskatchewan Cancer Agency, Saskatoon, Saskatchewan
- France (8):
  - Hopital Pontchaillou, Rennes, Brittany Region
  - Centre Hospitalier Universitaire de Limoges, Limoges, Limousin, Lorraine
  - Centre Hospitalier Universitaire Nantes - Hotel Dieu, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens, Picardie
  - Hopital Saint-Antoine, Paris, Île-de-France Region
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Île-de-France Region
  - Hopital Necker-Enfants Malades, Paris, Île-de-France Region
  - Hopital Saint Louis, Paris, Île-de-France Region
- Germany (7):
  - Universitatsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Diakonie-Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Universitatsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Universitatsklinikum Halle, Halle, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
- Greece (2):
  - University General Hospital of Athens Attikon, Athens, Attica
  - University Regional General Hospital of Patras, Patras, Peloponnese
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar, Hungary
- Israel (5):
  - Soroka University Medical Center, Beersheba, Beersheba
  - Rambam Health Care Campus - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Azienda Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria, Calabria
  - Azienda Ospedaliera Cardinale G. Panico, Tricase, Lecce
  - Ospedale Mazzoni, Ascoli Piceno, The Marches
  - Ospedale dell'Angelo, Mestre, Venezia
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Policlinico Universitario di Catania, Catania
  - Istituto Clinico Humanitas Humanitas Cancer Center, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Presidio Ospedaliero di Pescara, Pescara
- Japan (9):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Okayama University Hospital, Okayama, Okayama-ken
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-Ku, Tokyo
  - Osaka City University Hospital, Osaka
- Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico
- Oslo University Hospital - Rikshospitalet, Oslo, Norway
- Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship, Poland
- Portugal (3):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, Lisbon
  - Centro Hospitalar de Lisboa Norte EPE- Hospital Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, Porto
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Targu Mure, Târgu Mureş, Mureș County
  - Institutul Clinic Fundeni, Bucharest
- Russia (2):
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - National Research Center for Hematology, Moscow
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (11):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Keimyung University Dongsan Hospital, Daegu, Gyeongsangbuk-do
  - Pusan National University Hospital, Pusan, Gyeongsangnam-do
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus i Lund, Lund, Skåne County
  - Karolinska Universitetssjukhuset, Stockholm
- Switzerland (2):
  - Universitatsspital Basel, Basel
  - Universitatsspital Zurich, Zurich
- Taiwan (7):
  - Buddhist Tzu Chi General Hospital, Hualien City, Hualien
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (5):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, England
  - Barts Health NHS Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, England
  - Cardiff and Vale University Health Board, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Chen YB, Mohty M, Zeiser R, Teshima T, Jamy O, Maertens J, Purtill D, Chen J, Cao H, Rossiter G, Jansson J, Floisand Y. Vedolizumab for the prevention of intestinal acute GVHD after allogeneic hematopoietic stem cell transplantation: a randomized phase 3 trial. Nat Med. 2024 Aug;30(8):2277-2287. doi: 10.1038/s41591-024-03016-4. Epub 2024 Jun 6. PMID 38844797

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 95 investigative sites in Canada, United States, Argentina, Brazil, Belgium, France, Germany, Italy, Norway, Portugal, Spain, Sweden, Switzerland, United Kingdom, Austria, Greece, Hungary, Poland, Israel, Romania, Russia, Australia, Japan, Republic of Korea and Singapore from 6 February 2019 to 9 May 2022.
Pre-assignment Details: Participants undergoing allogeneic hematopoietic stem cell transplantation (Allo-HSCT) were randomized into 1:1 ratio to receive Vedolizumab 300 mg or vedolizumab-matching placebo. As pre-specified in the protocol, Day -1 corresponds to Day 1 of the ADaM data set, and similarly, Day 0 corresponds to Day 2. Therefore, the total duration becomes Day 182.
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, IV, once on Day -1 along with background graft-versus-host disease (GvHD) prophylaxis regimen prior to Allo-HSCT and once on Days +13, +41, +69, +97, +125, and +153 post Allo-HSCT up to the end of study treatment (up to 182 days).
Period: Overall Study
Arm/Group | Placebo | Vedolizumab 300 mg
Started | 169 | 174
Safety Analysis Set (Safety Analysis Set included all participants who received at least 1 dose of study drug.) | 165 | 169
Full Analysis Set (Full Analysis Set included all participants who were randomized, received at least 1 dose of the treatment, and under-went allo-HSCT.) | 165 | 168
Completed (Participants who completed the 182 days treatment period and the long term follow-up (6 months after the last dose of study drug).) | 98 | 117
Not Completed | 71 | 57
Not completed — Adverse Event | 5 | 6
Not completed — Protocol Deviation | 3 | 0
Not completed — Withdrawal by Subject | 18 | 16
Not completed — Site Termination | 1 | 0
Not completed — Unsatisfactory Therapeutic Response | 5 | 3
Not completed — Death | 33 | 26
Not completed — Death (COVID-19-Related) | 1 | 0
Not completed — Reason Not Specified | 5 | 5
Not completed — Other (COVID-19-Related) | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized, received at least 1 dose of the treatment, and under-went allo-HSCT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vedolizumab 300 mg | Total
Number analyzed (Participants) | 165 | 168 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (14.49) | 50.8 (14.41) | 51.4 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 103 | 209
  Male | 59 | 65 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 133 | 133 | 266
  Unknown or Not Reported | 23 | 19 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 29 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 114 | 121 | 235
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Intestinal aGvHD-Free Survival After Allo-HSCT by +180 Days
Description: Intestinal aGvHD Free Survival is the time from the date of first study drug administration (Day-1) to intestinal aGvHD event/death, where an event is defined as death due to any cause or Stage 1-4 intestinal involvement per Acute Graft versus-Host Disease Clinical Stage criteria. Data was censored for participants who have not had the intestinal aGvHD event or died or have had the event after pre-specified timing, e.g., last contact or Day +180 after allo HSCT whichever occurs first.
Time Frame: From the date of first dose of study drug to first documented intestinal aGvHD or death, whichever occurs first up to +180 days
Population: FAS included all participants who were randomized, received at least 1 dose of the treatment, and under-went allo HSCT. As pre-specified in the protocol, Day -1 corresponds to Day 1 of the ADaM data set, and similarly, Day 0 corresponds to Day 2. Therefore, the total duration becomes Day 182.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [14 to 182] — The median was not estimable due to censoring of participants. | NA [2 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.27 to 0.73]

2. Secondary Outcome: Intestinal aGvHD-Free and Relapse-Free Survival
Description: Intestinal aGvHD and Relapse Free Survival is the time from the date of first study drug administration (Day-1) to intestinal aGvHD event/death/relapse, where an event is defined as death or Stage 1-4 intestinal involvement per Acute Graft versus-Host Disease Clinical Stage criteria, or relapse. It will be censored for participants who have not had the event or have had the event after pre-specified timing, e.g., last contact or Day +180 after allo-HSCT whichever occurs first.
Time Frame: From the date of first dose of study drug to first documented intestinal aGvHD, death or relapse, whichever occurs first up to Day +180
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Groups:
- Placebo: Vedolizumab placebo-matching, IV infusion, once on Day -1 along with background GvHD prophylaxis regimen prior to Allo-HSCT and once on Days +13, +41, +69, +97, +125, and +153 post Allo-HSCT up to the end of study treatment (up to 182 days).
- Vedolizumab 300 mg: Vedolizumab 300 mg, IV, once on Day -1 along with background GvHD prophylaxis regimen prior to Allo-HSCT and once on Days +13, +41, +69, +97, +125, and +153 post Allo-HSCT up to the end of study treatment (up to 182 days).
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [14 to 182] — The median was not estimable due to censoring of participants. | NA [2 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p = 0.0043, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.37 to 0.86]

3. Secondary Outcome: Grade C-D aGvHD-Free Survival
Description: Grade C-D aGvHD Free Survival is the time from the date of first study drug administration (Day-1) to GvHD event/death, where an event is defined as Grade C-D aGvHD any organ involvement per International Bone Marrow Transplant Registry Database (IBMTR) Severity Index for aGvHD or death. It will be censored for participants who have not had the event or have had the event after pre-specified timing, eg, last contact or Day +180 after allo-HSCT whichever occurs first.
Time Frame: From the date of first dose of study drug to first documented Grade C-D aGvHD or death, whichever occurs first up to Day +180
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [12 to 182] — The median was not estimable due to censoring of participants. | NA [12 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p = 0.0204, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.39 to 0.91]

4. Secondary Outcome: Nonrelapse Mortality (NRM)
Description: Non-relapse mortality is the time from the date of first study drug administration (Day-1) to death without occurrence of a relapse. Data was censored for participants who have not had the event or have had the event after pre-specified timing, e.g., last contact or Day +180 after allo HSCT whichever occurs first.
Time Frame: From the date of first dose of study drug to first documented death without relapse, up to Day +180
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [14 to 182] — The median was not estimable due to censoring of participants. | NA [19 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p = 0.0668, Log Rank; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.22 to 1.04]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival by Days +180 is the time from the date of first study drug administration (Day-1) to death from any cause.
Time Frame: From the date of first dose of study drug to first documented death up to Day +180
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [14 to 182] — The median was not estimable due to censoring of participants. | NA [19 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p = 0.1458, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.34 to 1.17]

6. Secondary Outcome: Grade B-D aGvHD-Free Survival
Description: Grade B-D aGvHD Free Survival is the time from the date of first study drug administration (Day-1) to aGvHD event or death, where an event is defined as death or grade B-D any organ involvement per IBMTR Severity Index for aGvHD.
Time Frame: From the date of first dose of study drug to first documented grade B-D aGvHD or death, whichever occurs first up to Day +180
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Vedolizumab 300 mg
Number analyzed (Participants) | 165 | 168
days | NA [12 to 182] — The median was not estimable due to censoring of participants. | NA [12 to 182] — The median was not estimable due to censoring of participants.
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab 300 mg; Test type: Superiority; p = 0.0105, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.46 to 0.91]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to end of study (up to 39 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. All-cause mortality was collected for all enrolled participants. SAEs and Non-SAEs were collected for safety population. Safety Population included all participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 34/169 | 26/174
Serious Adverse Events (participants affected / at risk) | 114/165 | 120/169
Other Adverse Events (participants affected / at risk) | 164/165 | 169/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Vedolizumab 300 mg (N=169)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukopenias (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failures (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 13 | 13
Multiple organ dysfunction syndrome (General disorders) | 3 | 5
Disease progression (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Polyserositis (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Perforated ulcer (General disorders) | 1 | 0
Choleostasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 16 | 6
Acute graft versus host disease (Immune system disorders) | 5 | 2
Acute graft versus host disease in liver (Immune system disorders) | 2 | 5
Acute graft versus host disease in skin (Immune system disorders) | 4 | 3
Chronic graft versus host disease (Immune system disorders) | 1 | 2
Engraftment syndrome (Immune system disorders) | 2 | 1
Chronic graft versus host disease in liver (Immune system disorders) | 2 | 0
Graft versus host disease in eye (Immune system disorders) | 1 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 1
Acute graft versus host disease oral (Immune system disorders) | 1 | 0
Chronic graft versus host disease in lung (Immune system disorders) | 0 | 1
Chronic graft versus host disease in skin (Immune system disorders) | 0 | 1
Chronic graft versus host disease oral (Immune system disorders) | 1 | 0
Graft versus host disease in lung (Immune system disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Atypical mycobacterial infection (Infections and infestations) | 1 | 0
Acinetobacter infection (Infections and infestations) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 1 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 6
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Sinusitis fungal (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Human herpesvirus 6 encephalitis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 5
Tracheobronchitis (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 1 | 0
Human polyomavirus infection (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 9 | 4
Septic shock (Infections and infestations) | 4 | 4
Bacteraemia (Infections and infestations) | 5 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 1 | 0
Septic encephalopathy (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vascular device infection (Infections and infestations) | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Prescribed overdose (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Engraft failure (Injury, poisoning and procedural complications) | 0 | 4
Transplant failure (Injury, poisoning and procedural complications) | 1 | 3
Delayed engraftment (Injury, poisoning and procedural complications) | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1
Blast cell count increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 9
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Minimal residual disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Philadelphia positive acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 9
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hemorrhage intracranial (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 3
Mental status changes (Psychiatric disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 4
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 3
Renal failure (Renal and urinary disorders) | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiolitis obliterans syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=165) | Vedolizumab 300 mg (N=169)
Diarrhoea (Gastrointestinal disorders) | 102 | 95
Stomatitis (Gastrointestinal disorders) | 90 | 90
Nausea (Gastrointestinal disorders) | 83 | 85
Pyrexia (General disorders) | 62 | 80
Anaemia (Blood and lymphatic system disorders) | 72 | 68
Acute Graft Versus Host Disease in Skin (Immune system disorders) | 65 | 67
Febrile Neutropenia (Blood and lymphatic system disorders) | 54 | 67
Headache (Nervous system disorders) | 58 | 58
Hypomagnesaemia (Metabolism and nutrition disorders) | 52 | 60
Hypertension (Vascular disorders) | 54 | 54
Hypokalaemia (Metabolism and nutrition disorders) | 54 | 47
Vomiting (Gastrointestinal disorders) | 55 | 41
Constipation (Gastrointestinal disorders) | 47 | 43
Fatigue (General disorders) | 50 | 38
Decreased Appetite (Metabolism and nutrition disorders) | 40 | 45
Platelet Count Decreased (Investigations) | 47 | 38
Rash (Skin and subcutaneous tissue disorders) | 36 | 43
Thrombocytopenia (Blood and lymphatic system disorders) | 31 | 43
Neutropenia (Blood and lymphatic system disorders) | 32 | 40
Abdominal Pain (Gastrointestinal disorders) | 35 | 34
Insomnia (Psychiatric disorders) | 32 | 35
Cytomegalovirus Infection Reactivation (Infections and infestations) | 28 | 37
Oedema Peripheral (General disorders) | 35 | 29
Alanine Aminotransferase Increased (Investigations) | 26 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 28
Blood Creatinine Increased (Investigations) | 35 | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 36
Aspartate Aminotransferase Increased (Investigations) | 25 | 30
Dry Eye (Eye disorders) | 21 | 34
Dry Mouth (Gastrointestinal disorders) | 28 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 26
Blood Bilirubin Increased (Investigations) | 27 | 21
Dry Skin (Skin and subcutaneous tissue disorders) | 22 | 23
Dizziness (Nervous system disorders) | 23 | 21
Dysgeusia (Nervous system disorders) | 21 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 24
Acute Kidney Injury (Renal and urinary disorders) | 20 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 19
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 | 25
Tremor (Nervous system disorders) | 21 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (17) | 22 (23)
Erythema (Skin and subcutaneous tissue disorders) | 13 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 | 17
Dyspepsia (Gastrointestinal disorders) | 20 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 18 | 15
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 16 | 17
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 15 | 18
Abdominal Pain Upper (Gastrointestinal disorders) | 16 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 18
Blood Alkaline Phosphatase Increased (Investigations) | 15 | 16
Hypotension (Vascular disorders) | 12 | 19
Anxiety (Psychiatric disorders) | 14 | 14
Neutrophil Count Decreased (Investigations) | 15 | 13
White Blood Cell Count Decreased (Investigations) | 18 | 10
Asthenia (General disorders) | 12 | 14
Acute Graft Versus Host Disease In Intestine (Immune system disorders) | 15 | 10
Dysuria (Renal and urinary disorders) | 12 | 13
Abdominal Distension (Gastrointestinal disorders) | 11 | 13
Chronic Graft Versus Host Disease Oral (Immune system disorders) | 10 | 14
Proctalgia (Gastrointestinal disorders) | 15 | 9
Chronic Graft Versus Host Disease In Skin (Immune system disorders) | 7 | 16
Chronic Graft Versus Host Disease (Immune system disorders) | 12 | 10
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Haematuria (Renal and urinary disorders) | 13 | 9
Haemorrhoids (Gastrointestinal disorders) | 8 | 14
Chills (General disorders) | 10 | 11
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 12 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Vision Blurred (Eye disorders) | 11 | 10
Oedema (General disorders) | 13 | 7
Depression (Psychiatric disorders) | 6 | 13
Neuropathy Peripheral (Nervous system disorders) | 9 | 10
Oral Pain (Gastrointestinal disorders) | 7 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7) | 12 (12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 7 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9)
Tachycardia (Cardiac disorders) | 6 (9) | 12 (13)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 8 (9)
Hypervolaemia (Metabolism and nutrition disorders) | 9 (11) | 7 (8)
Pollakiuria (Renal and urinary disorders) | 7 (8) | 9 (9)
Pain (General disorders) | 11 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Flatulence (Gastrointestinal disorders) | 10 | 4
Confusional State (Psychiatric disorders) | 10 | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 9
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03657160/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT03657160/SAP_001.pdf